CLINICAL TRIAL: NCT03835754
Title: Heart Expand Continued Access Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-CAR-121918
Record Dates: First submitted 2019-01-22; First posted 2019-02-11 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2022-12

CONDITIONS: Heart Transplant
Keywords: Heart preservation; Beating heart transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- OCS Preservation (Experimental)
  Interventions: Device: OCS Heart System

INTERVENTIONS:
Device: OCS Heart System — The OCS Heart System preserves the heart in a near-physiological, beating state by perfusing the heart with a warmed, donor-blood based perfusate that is supplemented with nutrients and oxygen in a controlled and protected environment

SUMMARY:
The OCS™ Heart System will be used to preserve and assess donor hearts that do not meet current standard donor heart acceptance criteria for transplantation in this continued access protocol.

DETAILED DESCRIPTION:
To provide additional data evaluating the safety and effectiveness of the OCS™ Heart System to preserve and assess donor hearts that do not meet current standard donor heart acceptance criteria (as identified above) for transplantation to potentially improve donor heart utilization for transplantation at a range of transplant centers in the U.S. and to permit patients and physicians access to the OCS Heart System while a PMA application is under preparation and review.

ELIGIBILITY:
Inclusion Criteria (DONOR):

At least one of the following:

* Expected total cross-clamp time of ≥ 4 hours
* Expected total cross-clamp time of ≥ 2 hours PLUS one or more of the following risk factors Donor age 45-55 years, inclusive, with no coronary catheterization data; or Donor age ≥ 55 years; or Left ventricular septal or posterior wall thickness of >12 mm, but ≤ 16 mm; or Reported down time of ≥ 20 min, with stable hemodynamics at time of final assessment; or Left heart ejection fraction (EF) ≥ 40%, but ≤ 50% at time of acceptance of offer; or Donor angiogram with luminal irregularities with no significant CAD (≤ 50%); or History of carbon monoxide poisoning with good cardiac function at time of donor assessment; or Social history of alcoholism with good cardiac function at time of donor assessment; or History of diabetes without significant CAD (≤ 50%) on angiogram.

Exclusion

* CAD with > 50% stenosis on angiogram, or
* Cardiogenic shock or myocardial infarction, or
* EF consistently < 40%, or
* Significant valve disease except for competent bicuspid aortic valve.

Eligibility Criteria (RECIPIENT)

* Registered primary heart transplant candidate
* Age >18 years old
* Written informed consent. Exclusion
* Prior solid organ or bone marrow transplant
* Chronic use of hemodialysis or renal replacement therapy for diagnosis of chronic renal insufficiency requiring dialysis
* Multi-organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Cedars-Sinai, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - AdventHealth Orlando, Orlando, Florida
  - St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Nyph/Cumc, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Schroder JN, Patel CB, DeVore AD, Casalinova S, Koomalsingh KJ, Shah AS, Anyanwu AC, D'Alessandro DA, Mudy K, Sun B, Strueber M, Khaghani A, Shudo Y, Esmailian F, Liao K, Pagani FD, Silvestry S, Wang IW, Salerno CT, Absi TS, Madsen JC, Mancini D, Fiedler AG, Milano CA, Smith JW. Increasing Utilization of Extended Criteria Donor Hearts for Transplantation: The OCS Heart EXPAND Trial. JACC Heart Fail. 2024 Mar;12(3):438-447. doi: 10.1016/j.jchf.2023.11.015. Epub 2024 Jan 24. PMID 38276933

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCS Preservation
Started | 75
Completed (Completed one-year follow-up) | 71
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | OCS Preservation
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival at Day 30 Post-transplantation and Absence of Severe PGD (Left or Right Ventricle) in the First 24 Hours Post-transplantation
Description: A composite of patient survival at Day 30 and absence of severe primary heart graft dysfunction (PGD) (LV or RV) in the first 24 hours post-transplantation according to ISHLT consensus manuscript in the protocol.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preservation
Number analyzed (Participants) | 75
Participants | 72
Statistical Analysis 1: Comparison: OCS Preservation; Test type: Other — Confidence internal is 88.8%, upper bound limit 99.2%; Clopper Pearson exact confidence interva = 96, 95% CI 2-sided [88.8 to 99.2]

ADVERSE EVENTS:
Time Frame: Per the protocol, all SAEs and heart graft related SAEs will be collected for the first 30 days post-transplant. All-Cause Mortality was assessed for 12 months post-transplant as reported.
Description: Per the protocol, only serious adverse events (SAEs) and Heart Graft-Related SAE's (HGRSAEs) will be captured in this study.
  Not Serious AEs were not collected, and therefore not reported.
Arm/Group | OCS Preservation
All-Cause Mortality (participants affected / at risk) | 71/75
Serious Adverse Events (participants affected / at risk) | 44/75
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Preservation (N=75)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 5 (5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 6 (6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Acute cellular rejection (Immune system disorders) | 3 (3)
Acute graft rejection (Immune system disorders) | 3 (3)
Bacteremia (Infections and infestations) | 2 (2)
Escherichia coli infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 (1)
Injury to inferior vena cava (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Volume overload (Metabolism and nutrition disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Hemorrhagic stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Nerve pain (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Psychosis (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 10 (10)
Acute tubular necrosis (Renal and urinary disorders) | 1 (1)
Kidney dysfunction (Renal and urinary disorders) | 2 (2)
Bronchial mucus plug (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Bleeding (Vascular disorders) | 8 (8)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT03835754/Prot_SAP_000.pdf